CLINICAL TRIAL: NCT02180620
Title: Exercise Timing and Postprandial Glycemia in Type 2 Diabetes
Brief Title: Pre-dinner vs. Post-dinner Exercise on Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: exertime
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes
Keywords: GIP; GLP-1; exercise timing; resistance exercise; glucose concentrations
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No exercise (Experimental): participants will remain sedentary during testing
  Interventions: Other: No exercise
- Meal then exercise (Experimental): 45 min of resistance training will be performed after a standard meal
  Interventions: Other: Meal then exercise
- exercise then meal (Experimental): 45 min of resistance training will be performed prior to a standard meal
  Interventions: Other: exercise then meal

INTERVENTIONS:
Other: No exercise — During the no exercise trial (NoEX), the participants will remain sedentary during testing.
  Other Names: NoEX
  Arms: No exercise
Other: Meal then exercise — During the post-meal exercise trial (M→EX), 45 min of resistance training will be performed
  Other Names: M-EX
  Arms: Meal then exercise
Other: exercise then meal — During the exercise prior to the meal trial (EX→M), 45 min of resistance training will be performed
  Other Names: EX-M
  Arms: exercise then meal

SUMMARY:
With many medications we prescribe them relative to time of day or a meal. This study established if pre dinner vs post dinner exercise was more effective at altering post dinner glucose and triglyceride levels vs no exercise at all.

DETAILED DESCRIPTION:
All participants completed three trials in a random order in which they consumed a standardized dinner meal with 1) no RE (NoRE), 2) pre-dinner RE (RE→M), and 3) post-dinner RE beginning 45 min after dinner (M→RE). Diet was standardized during the day of testing. Participants reported to the lab for testing sometime between 3 - 5:30 p.m. and upon arrival a venous catheter was inserted into a forearm vein. Frequent blood sampling, indirect calorimetry measurements, and subjective well-being measurements ensued for ~5.75 h while the participants were in the lab.

ELIGIBILITY:
Inclusion Criteria:

* Obese ( body mass index 30-45 kg/m2)
* Physician diagnosed with type 2 diabetes receiving standard medical care
* Non-smokers
* Pregnancy
* Lactating mothers

Exclusion Criteria:

* Insulin
* Surgical weight loss
* Orthopedic limitations to exercise
* Weight loss in the previous 3 months

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
glucose concentrations | Blood samples were taken every 5-10 min during the first 3.7 h of testing and every 30 min during the last 2 h

SECONDARY OUTCOMES:
triglyceride concentrations | Blood samples were taken every 5-10 min during the first 3.7 h of testing and every 30 min during the last 2 h

OTHER OUTCOMES:
GLP-1 concentrations | Blood samples were taken every 5-10 min during the first 3.7 h of testing and every 30 min during the last 2 h

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heden TD, Liu Y, Kanaley JA. A comparison of adipose tissue interstitial glucose and venous blood glucose during postprandial resistance exercise in patients with type 2 diabetes. J Appl Physiol (1985). 2018 Apr 1;124(4):1054-1061. doi: 10.1152/japplphysiol.00475.2017. Epub 2017 Sep 28. PMID 28970202